CLINICAL TRIAL: NCT01713010
Title: Evaluation of Integrated Predictive Index of Weaning From Mechanical Ventilation in Patients With Traumatic Brain Injury
Brief Title: Study of Variables Related to the Discontinuation of Mechanical Ventilation in Patients With Head Injury
Acronym: INDEXTBI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, Camila Marques Dias, Physiotherapist, Federal University of Uberlandia
Other Study IDs: 11212PSC002
Record Dates: First submitted 2012-10-22; First posted 2012-10-24 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Traumatic Brain Injury; Weaning Failure; Mechanical Ventilation Complication
Keywords: Keywords provided by Atlantic Health System:; Rapid Shallow Breathing Index; Mechanical Ventilation; Additional relevant MeSH terms:; Respiration Disorders; Traumatic Brain Injury; Weaning Failure; Mechanical ventilation complication
MeSH Terms: conditions — Brain Injuries, Traumatic; Respiration Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Predictive indexes of weaning from mechanical ventilation
  Other Names: respiratory frequency to tidal volume (f/VT); airway occlusion pressure(P0.1)

SUMMARY:
The purpose of this study is to evaluate physiological variables to the decision about the appropriate time to discontinuation of mechanical ventilation in patients with traumatic brain injury. It is expected that these variables are effective in predicting the outcome of weaning from mechanical ventilation.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effectiveness of integrated pressure index of airway occlusion x index breathing fast and shallow (p 0.1 x f/VT) in predicting success and failure of weaning from mechanical ventilation in patients with traumatic brain injury.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic Brain Injury (TBI)
* Patients using artificial airway (intubation and / or tracheostomy)
* Recovery from the acute phase of the disease underlying
* Both sexes
* Ventilation mode pressure support (PSV), pressure support (PS) required to ensure a tidal volume (VT) = 6 to 8 ml / kg
* Age over 18 years
* Hemoglobin > 7 g/dL
* Duration of mechanical ventilation longer than 24 hours
* Body temperature < 38 degrees
* pH ≥ 7.30
* PaO2 ≥ 60 mmHg with FiO2 ≤ 0.4 and PEEP ≤ 8 cmH2O
* Glasgow Coma Scale ≥ 8 or tracheostomized
* Sedative agents minimum dosages to to maintain values of 2 or 3 on the Ramsay Scale

Exclusion Criteria:

* Admitted to the ICU with artificial airways held in other institutions
* Surgery scheduled for the next 72 hours
* Withdrawal of consent from parents at any stage of the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the intensive care unit with brain trauma in the process of weaning from mechanical ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2012-03; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Result weaning mechanical ventilation in patients with traumatic brain injury,analyzing success and failure of weaning by 0.1 p and f / VT. | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Camila Marques Dias, Principal Investigator — Federal University of Uberlandia; Célia Regina Lopes, Study Chair — Federal University of Uberlandia
Locations (1):
- Federal University of Uberlandia, Uberlândia, Minas Gerais, Brazil